CLINICAL TRIAL: NCT05381610
Title: A Clinical Investigation Evaluating Peristeen® Performance Characteristics of Scintigraphic Measurements in Patients With Neurogenic Bowel Dysfunction
Brief Title: A Clinical Investigation Evaluating Peristeen® Performance
Acronym: CP342
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment - Sponsor decision
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP342
Record Dates: First submitted 2022-03-14; First posted 2022-05-19 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-04

CONDITIONS: Neurogenic Bowel
MeSH Terms: conditions — Neurogenic Bowel

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neurogenic Bowel (Experimental): This is a US-Only, early feasibility, Investigational Device Exemption - Non-Significant Risk (IDE-NSR), single-center, open label study evaluating the effects of Peristeen, compared to a LVE administered into the rectum. The subjects to be analysed will be subjects with : Neurogenic Bowel Dysfunction (NBD). The NBD cohort will be broken down into two phases: LVE and Peristeen. See Statistical section 10 for more infor-mation on cohort and sub-group analyses.
  Interventions: Device: Peristeen

INTERVENTIONS:
Device: Peristeen — The Peristeen system will be handled by Coloplast trained personnel. The investigator and a trained nurse will participate in all the investigation related procedures. The nurse is trained in the handling of the investi-gational product as well as this is described in detail in the Instruction for Use (IFU). Subjects (and their caregivers, if appropriate) will also be trained on the use of Peristeen prior to independent use at home.

SUMMARY:
Peristeen has been on the market globally since 2006 and marketed in the US since 2012, and more than 10,000 patients worldwide have been using Peristeen, with over 3,000 patients in the US. However, the US reimbursement is not uniform, resulting in many patients suffering from NBD in sub-optimal bowel manage-ment. Therefore, this study will scientifically define and describe how the Peristeen system is different from a large volume enema.

DETAILED DESCRIPTION:
The Peristeen system is a non-surgical, FDA-cleared, Class II device for the treatment of patients with neu-rogenic bowel dysfunction (NBD) who have failed conservative bowel management treatment and would otherwise be considered candidates for surgery. (Note: The Peristeen pump with connectors and tubing only is considered to be a FDA class I device. When associated with the rectal balloon catheters, the Peristeen system is considered a class II device thereby giving the entire System an overall designation of class II.) The Peristeen system is a non-surgical, manual system, consisting of a control unit (featuring a pneumatic bulb pump and a four-position rotary switch), a water bag (featuring a pressure relief valve), tubes and con-nectors up to a lubricated catheter which is inserted into the anal canal to allow water to enter the bowel. The system is also accompanied by straps to secure the system on the thigh while being used. The Peristeen catheter is equipped with a balloon which may be inflated or deflated with air once positioned in the rectum. Peristeen has been on the market globally since 2006 and marketed in the US since 2012. More than 10,000 patients worldwide have been using Peristeen, with over 3,000 patients in the U.S (United States).

Neurogenic Bowel Dysfunction (NBD) as defined by the American Academy of Physical Medicine and Re-habilitation, is an, "impairment of the gastrointestinal and anorectal function from a lesion in the nervous system." These neurological lesions can come from a range of disease states, such as, but not limited to spina bifida, multiple sclerosis, Parkinson's, and Spinal Cord Injury (SCI) . Numerous publications and findings have been conducted in humans using Peristeen, with over 120 publications in just the past 5 years.

As a result of the inability to evacuate the bowel, NBD patients experience fecal constipation, fecal impaction, and/or a failure to contain stool in the bowel (i.e., fecal incontinence). These defecation disturbances can be severe enough that they can increase a patient's risk for repeated emergency care. The prevalence of NBD is well documented and occurs in both children and adults. For example, not only do these constipation issues prevail in children and young adults with spina bifida, approximately one third of the NBD patients are fecally incontinent. These resulting complications with bowel management results in an increased risk for urinary tract infections (UTIs), due to the anatomical proximity of the bowel and lower urinary tract. Specific to SCI patients, literature reports that 95% require more than one intervention to initiate defecation.

Quality of life for this patient population has been observed to decline as the severity of NBD increases and patients with SCI report that bowel dysfunction has a greater negative impact on life than any other SCI-related impairment with approximately 50% reporting moderate-to-severe NBD symptoms. The symptoms of NBD and the inability to management their bowels can cause significant emotional distress, affecting self-esteem, personal relationships, and social life.

The time required for bowel management is also a factor of a NBD patient's life. Many patients with NBD spend a significant part of their day on bowel management with 14% to 63% spending more than 1 hour on each episode. Furthermore, complete assistance from a care giver is required by 23% and some help is required by 12%. Peristeen's ergonomic design, leg strap, pump mechanism, inflatable balloon, makes it possible for immobilized patients or those with poor hand function to conduct the procedure them-selves, thereby allowing for personal independence and privacy/discreteness.

Peristeen is differentiated from standard bowel care and its clinical superiority and cost-effectiveness have been clearly demonstrated in patients with NBD. An analysis of real-life data in N = 227 NBD patients who have failed standard bowel care (SBC) and has found that Peristeen can reduce the stoma surgery rate by 64% in the first 2 years after treatment initiation and 35% over a lifetime. Specifically, the 2-year stoma surgery rate for Peristeen vs. standard bowel care is 2% vs. 6%, respectively. Furthermore, in a human clinical trial, N = 49; MS patients showed a decrease in hospitalizations of 41% per year when patients use Peristeen. Without Peristeen, the physical issues that arise result in an increase in healthcare utilization. For example, adults with NBD have been shown to be more than twice as likely to be admitted to the hospital due to fecal impaction and constipation in comparison to healthy individuals. If not managed properly, NBD can ultimately lead to stoma surgery or need for permanent residential care.

Despite the documented clinical success with Peristeen, it is marginally accessible due in large part to a misclassification as a large volume enema (LVE). Typically, LVE is an over-the-counter product that consists of a water bag or bladder, tubing with adjustable clamp to connect and start/stop the gravity-fed water flow to the rectal catheters/probe, and a hook or ability to hang the bag. As gravity is used to administer and adjust the flow of water into the rectum, the patient typically needs assistance and/or needs to lay on the floor near the toilet to administer. Peristeen has an adjustable/inflatable balloon catheter to allow for a complete seal in the rectum where LVEs do not, thereby allowing patients to sit on the toilet or commode during the process. The leg strap and ergonomic dial and pump also allow the patient to perform the procedure independently.

Treatments like LVE are noted to be difficult to retain fluid in patients as there is no secure way to seal the rectum, thus much of the fluid involuntarily flowing out during installation. In addition, published literature characterizing the quantity of fecal removal with LVE is lacking and is an uncommon use in practice, thus, there is no understanding of how well they fully empty the colon. In Spinal Cord Injury patients, bowel distension caused by LVEs has been reported to trigger autonomic dysreflexia. Thus, the purpose of this study will be to investigate and compare the effects of both a large-volume enema and Peristeen on emptying of the colon.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be diagnosed with neurogenic bowel dysfunction (NBD), plus:

   * Neurogenic bowel dysfunction score (Appendix A) of 10 or higher, indicating moderate or severe NBD AND
   * Documented failure to achieve adequate bowel management in the last 30-days using the standards of care regimen including medications that alter GI transit but is naïve* to LVE and Peristeen

   NOTE: For this study only, subjects are required to be naive for statistical analyses purposes.

   For Spinal Cord Injury Subjects Only: Is past or outside initial spinal cord shock window
3. Be at least 18 years of age and have full legal capacity
4. Be willing and able to comply with investigation procedures - includes ability to forgo any rectal stimulation, rectal therapies or rectally administered medications or treatments for the duration of the study
5. Have a normal digital examination on file in the past 6 months.
6. Anorectal manometry test and data on file within past 6 months.
7. Successful balloon expulsion test on file within the past 6 months. (i.e., can expel the balloon in 120 seconds or less)
8. In the opinion of the investigator, be an appropriate candidate for the study

Exclusion Criteria:

1. Have history/episode of severe autonomic dysreflexia, bradycardia or tachycardia.
2. History of bowel perforation
3. Have known anal or colorectal stenosis
4. Have active/recurrent colorectal cancer
5. Have active inflammatory bowel disease and/or Crohn's disease
6. Any of the following anal conditions: Anal fissure, anal fistula or third- or fourth-degree haemorrhoids
7. Have any history of irradiation therapy or chemotherapy targeting the abdomen and/or pelvic region
8. Have any history of gastrointestinal, anal, and/or colorectal surgery (i.e., appendectomy, tubal ligation or hysterectomy, hemorrhoidectomy, cholecystectomy, and/or hiatal hernia surgery, LARS, MACE)
9. Be within 4 weeks of endoscopic polypectomy (includes biopsy and/or endoscopy)
10. Have an implanted stimulation device of any kind.
11. Have ischemic colitis
12. Have chronic or complex diverticular disease (i.e., acute, severe, ulcerative, previous and/or abscess)
13. Have history of colonic obstruction, structural diseases of the colon or ileus
14. Are pregnant, planning on becoming pregnant, or breastfeeding
15. Have known phthalate sensitivity, specifically dibutyl phthalate
16. Are current user of Peristeen or Large Volume Enemas
17. Chronically used Peristeen or Large Volume Enema in the past 2 years.
18. Diagnosis of opioid-induced constipation and/or narcotic bowel syndrome.
19. Have severe Cognitive or severe physical impairment that prevents the ability to administer Peristeen by themselves and/or lack of caregiver support to administer Peristeen administration.
20. Have other individual factors, in the opinion of the physician/healthcare professional, in which participating is contraindicated.
21. Participation in concomitant clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
The differences in the scintigraphy images, i.e. percentage of fecal matter, will be compared between the LVE and Peristeen. | 72 days
  The subject's fecal matter movement will be measured radiologically and the percent changes in both a large-volume enema and Peristeen treatment will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No